CLINICAL TRIAL: NCT00617578
Title: Fast VT Episodes Are Terminated by ATP One Shot
Acronym: FavoriteATP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA080
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2012-05

CONDITIONS: Ventricular Tachycardia, Monomorphic
Keywords: Antitachy pacing; Implantable cardioverter-defibrillator
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): programming of VF therapy: ATP (antitachycardia pacing) One Shot ON
  Interventions: Device: ATP One Shot ON
- 2 (Active Comparator): programming of VF therapy: ATP (antitachycardia pacing) One Shot OFF
  Interventions: Device: ATP One Shot OFF

INTERVENTIONS:
Device: ATP One Shot ON — The new antitachycardia pacing algorithm "ATP One Shot" attempts to terminate fast VT by one ATP sequence and thus avoid defibrillation shock delivery
  Arms: 1
Device: ATP One Shot OFF — Standard defibrillation shock delivery
  Arms: 2

SUMMARY:
Many arrhythmias detected in the ventricular fibrillation (VF)-zone picture monomorphic ventricular tachycardia (VT) and, hence, could be terminated by antitachycardia pacing (ATP) treatment. Advantages of successful ATP are the painlessness termination and the shortened duration of arrhythmia. The ATP One Shot algorithm is integrated in the latest family of implantable cardioverter defibrillators (ICDs) from BIOTRONIK (Lumax). It allows a single delivery of ATP before charging capacitors to terminate lethal arrhythmia by painful shock.

The present study evaluates the efficacy of the ATP One Shot algorithm for the termination of fast VT episodes. 200 patients with secondary prophylactic ICD indication will be followed for 18 months. Spontaneous episodes detected in the VF-zone of the ICD will be evaluated with regard to cycle length, episode duration and course of device therapy.

DETAILED DESCRIPTION:
ICDs provide different detection zones for the therapy of VT and VF. An established form of therapy in the VT-zone is antitachycardia pacing (ATP). It is an effective, safe and painless method to terminate episodes of slow VT with a cycle length > 300 ms. Episodes detected in the VF zone will result in the delivery of a high-energy shock to terminate life-threatening VF. Many arrhythmia detected in the VF-zone picture monomorphic VT and could be easily terminated by ATP. Advantages of a successful termination by ATP therapy would be the painlessness and the shortened duration of the episode, as there would be no need to load shock capacitors. Fast VT are often hemodynamically poorly tolerated by the patient and should be terminated within very short time. The ATP One Shot algorithm is integrated in the latest family of ICDs from BIOTRONIK (Lumax) to allow a single delivery of ATP before charging capacitors.

The main objective of the study is the assessment of the efficacy of the ATP One Shot algorithm for the termination of fast VT episodes. To this end, spontaneous episodes detected in the VF-zone of the ICD are evaluated with regard to cycle length, episode duration and course of device therapy. In the context of the study, a confirmatory (hypothesis-testing) primary problem is investigated. The goal is to measure the time to first adequate shock therapy for episodes detected in the VF-zone of the device and to analyze the hazard ratio of the standard ICD setting compared to a therapy with the ATP One Shot algorithm.

The clinical project is conducted as randomized prospective multicenter study. The chronological order and the scope of the follow-ups meet the medical standard according to the international guidelines. A center-based, stratified block randomization will be performed. In approximately 50% of the patients the ATP One Shot algorithm will be activated, while the other 50% will be randomized into the control group.

A total of about 20 European investigational sites will participate in the study. Each center should enroll about 10 patients who will be followed for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* ICD indication for reason of survived cardiac arrest, ventricular tachycardia or syncope

Exclusion Criteria:

* ICD indication for reason of non-sustained VT post MI, positive family history for SCD (Brugada-, long/short QT-Syndrome), hypertrophic cardiomyopathy, primary prophylactic indication (e.g. SCD-HeFT, Madit II)
* Patients not capable of participating in the follow-ups
* Minors and pregnant women
* Patients who are already enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2007-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Time to the first adequate device shock | 18 months

SECONDARY OUTCOMES:
Quality of Life | 18 months
Duration of Episodes | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Otto Schwab, PD Dr., Study Chair — University Hospital Bonn, Germany
Locations (14):
- Austria (3):
  - Medizinische Abteilung, LKH Bruck, Bruck / Mur
  - Innere Medizin - Kardiologie, Universitätsklinik Innsbruck, Innsbruck
  - Med. Abteilung, AKH Linz, Linz
- Cardiology, Satakunta Central Hospital, Pori, Finland
- Germany (9):
  - Klinik für Innere Medizin, Vivantes Humboldt Klinikum, Berlin
  - Medizinische Klinik II, Universitätsklinikum Bonn, Bonn
  - Medizinische Klinik I, Ev. Krankenhaus, Holzminden
  - Medizinische Klinik, Kreiskrankenhaus, Neustadt / Aisch
  - Kardiologie, DRK Krankenhaus Mölln, Ratzeburg
  - Kardiologische Praxis Dr. Placke, Rostock
  - Innere Medizin - Kardiologie, Klinikum Uckermark, Schwedt
  - Kliniken Villingen Schwenningen, Klinik für Innere Medizin III, Kardiologie, Villingen
  - Medizinische Klinik I, St-Josefs-Hospital, Wiesbaden
- Cardiology, Rabin MC, Petah Tikva, Israel